CLINICAL TRIAL: NCT02500680
Title: A Phase IA/IB Trial to Evaluate the Safety, Tolerance, and Immunogenicity of MAS-1-Adjuvanted Seasonal Inactivated Influenza Vaccine (MER4101) With Hemagglutinin Dose Escalation Compared to Non-Adjuvanted Comparator Inactivated Influenza Vaccine (IIV) Standard Dose (SD) in Healthy Adults and High Dose (HD) IIV in Ambulatory Elderly Subjects
Brief Title: The Safety, Tolerance, and Immunogenicity of MAS-1-Adjuvanted Seasonal Inactivated Influenza Vaccine (MER4101)
Acronym: MER4101
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nova Immunotherapeutics Limited (Industry)
Collaborators: Mercia Pharma Inc. (Industry); Nova Laboratories Limited (Industry); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MPE002
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Influenza, Human
Keywords: Influenza; Adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Group 1 (Phase 1A) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) 1µg (Standard Dose) Single Dose
  Interventions: Biological: MER4101
- Group 2 (Phase 1A) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) 3µg (Standard Dose) Single Dose
  Interventions: Biological: MER4101
- Group 3 (Phase 1A) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) 5µg (Standard Dose) Single Dose
  Interventions: Biological: MER4101
- Group 4 (Phase 1A) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) 9µg (Standard Dose) Single Dose
  Interventions: Biological: MER4101
- Group 5A (Phase 1A) (Active Comparator): Fluzone quadrivalent influenza vaccine (Sanofi Pasteur) 15µg (Standard Dose) Single Dose
  Interventions: Biological: Inactivated Influenza Vaccine
- Group 5B (Phase 1B) (Active Comparator): Fluzone quadrivalent influenza vaccine (Sanofi Pasteur) 60µg (High Dose) Single Dose
  Interventions: Biological: Inactivated Influenza Vaccine
- Group 6 (Phase 1B) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) Optimal Vaccine Dose from Phase 1A (9µg) (Standard Dose) Single Dose
  Interventions: Biological: MER4101
- Group 7A (Phase 1B extension) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) 9µg/HA in 0.5 mL MAS-1 emulsion (Standard Dose) Single Dose
  Interventions: Biological: MER4101
- Group 7B (Phase 1B extension) (Active Comparator): Fluzone quadrivalent influenza vaccine (Sanofi Pasteur) 60µg (High Dose) Single Dose
  Interventions: Biological: Inactivated Influenza Vaccine
- Group 8A (Phase 1B extension) (Experimental): MER4101 (MAS-1 Adjuvanted IIV [Fluzone quadrivalent influenza vaccine, Sanofi Pasteur]) 15µg/HA in 0.5 mL MAS-1 emulsion (Standard Dose) Single Dose (as 2 x 0.25 mL in each arm)
  Interventions: Biological: MER4101
- Group 8B (Phase 1B extension) (Active Comparator): Fluzone quadrivalent influenza vaccine (Sanofi Pasteur) 60µg (High Dose) Single Dose (0.5 mL) in one arm and 0.5 mL of PBS in the other arm
  Interventions: Biological: Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: MER4101
  Other Names: Inactivated Influenza Vaccine with MAS-1 Adjuvant
  Arms: Group 1 (Phase 1A); Group 2 (Phase 1A); Group 3 (Phase 1A); Group 4 (Phase 1A); Group 6 (Phase 1B); Group 7A (Phase 1B extension); Group 8A (Phase 1B extension)
Biological: Inactivated Influenza Vaccine — Fluzone quadrivalent Influenza Vaccine
  Arms: Group 5A (Phase 1A); Group 5B (Phase 1B); Group 7B (Phase 1B extension); Group 8B (Phase 1B extension)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance, and immunogenicity of MAS-1-Adjuvanted seasonal inactivated influenza vaccine (IIV) (MER4101) with hemagglutinin dose escalation compared to non-adjuvanted comparator IIV standard dose (SD) in healthy adults and high dose (HD) IIV in ambulatory elderly subjects.

Hypothesis: Reduced HA dose IIV formulated in MAS-1 adjuvant (MER4101) has been shown under Phase 1A to be safe, tolerable and demonstrated a more robust and durable immune response to IIV over 6 months post-vaccination in healthy young adults 18 - 49 years of age compared to SD IIV. Under phase 1B, the 9 µg/HA dose of IIV in 0.3 mL MAS-1 was safe and well tolerated and immunogenically comparable to or better than 60 µg/HA HD IIV control over 3 to 6 months post-vaccination than HD IIV control. It is anticipated that the increased total dose of 15 µg HA antigen administered concurrently to opposite arms in 2 doses of 7.5 µg/HA IIV in 0.25 mL MAS-1 adjuvant emulsion will be safe, well tolerated, and more immunogenic than 9 µg/HA IIV in MAS-1, and will be more immunogenic when compared to HD IIV control in adults who are 65 years of age and older with the potential to provide better protection throughout the influenza season.

DETAILED DESCRIPTION:
The study is a Phase 1A, 1B and 1B extension, randomized, double-blind, single-center, clinical trial, in healthy adults (18-49 years old) and ambulatory elderly subjects (aged 65 years and older). Phase IA evaluated the safety, tolerability and hemagglutination inhibition assay (HAI) antibody response to MER4101 at each of four escalating doses of seasonal inactivated influenza vaccine (IIV) hemagglutinin (HA) antigen with a fixed dose of a water-in-oil emulsion adjuvant MAS-1 (Mercia Adjuvant System-1), compared with licensed, unadjuvanted, standard dose (SD) of licensed inactivated trivalent influenza virus vaccine (IIV). Phase IB evaluated the optimal dose of IIV in MAS-1 selected under phase IA for safety, tolerability and HAI antibody response (from Phase 1A known to be 9 µg of HA antigen in 0.3 mL dose of MAS-1 adjuvanted emulsion) in ambulatory elderly subjects compared to high dose (HD) IIV. The Phase 1B extension will evaluate if the increased dose volume of MAS-1 (0.5 mL vs 0.3 mL) at the same 9 µg/HA adjuvanted IIV vaccine is safe, well tolerated and immunogenic, and then whether the increased dose of 15 µg/HA in 0.5 mL MAS-1 is safe, well tolerated and still more immunogenic in elderly subjects.

The ability of standard dose (SD) IIV to protect against seasonal influenza virus infection in the elderly is less than vaccine efficacy observed in healthy young adults. The MAS-1-adjuvanted influenza virus vaccine offers the potential for higher seroconversion and seroprotection rates, hemagglutination inhibition (HAI) antibody titers relative to pre-vaccination HAI titers (GMFI), hemagglutinin (HA) antigen dose-sparing and cross-protection against antigenically divergent viral strains, and importantly, prolonged duration of protective immunity lasting up to at least 6 months post-vaccination in both the general adult population and the elderly, thereby providing potentially protective immunity throughout the influenza season. This study will determine if the adjuvanted vaccine formulated with one or more of the reduced HA antigen doses is safe. The study will also determine if it is likely to induce an improved HA antibody response (HAI) when compared to SD IIV in healthy adults and HD IIV in elderly subjects. This trial will inform future clinical trials in at-risk populations of older patients.

ELIGIBILITY:
Inclusion Criteria:

Specifically Phase 1A:

1. Males or non-pregnant females, 18 to 49 years old, inclusive.
2. Female subjects of childbearing potential who must agree to practice avoidance of pregnancy, including use of acceptable forms of contraception.
3. Pulse is 55 to 100 bpm, inclusive.
4. Systolic blood pressure is 90 to 140 mmHg, inclusive.
5. Diastolic blood pressure is 55 to 90 mmHg, inclusive.

For Phase 1B and Phase 1B Extension:

1. Ambulatory persons aged at least 65 years or older on the day of enrollment. Subjects will be considered ambulatory if they are not institutionalized, bedridden, or homebound.
2. Pulse is 50 to 115 bpm, inclusive.
3. Systolic blood pressure is 85 to 160 mmHg, inclusive.
4. Diastolic blood pressure is 55 to 95 mmHg, inclusive.

For Phase 1A, Phase 1B, and Phase 1B Extension:

1. Written informed consent form and Authorization to Obtain and Release Protected Health Information (HIPAA) form signed, prior to initiation of any study procedures
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are in good health, as determined by vital signs, medical history, and physical examination based on medical history to ensure any existing medical diagnoses or conditions are stable.
4. Stable chronic medical condition
5. Oral temperature is less than 100.4°F
6. Within institutional normal ranges for safety labs
7. Have a Body Mass Index (BMI) of 18-35

Exclusion Criteria:

Specifically Phase 1A:

1. Female subjects who are breastfeeding or plan to breastfeed at any given time from the study vaccination until 30 days after the study vaccination will be ineligible
2. Receipt of 2014-2015 and 2015-2016 seasonal influenza vaccine.
3. After 03 September 2015, any subject who intends to receive the 2015-2016 licensed influenza vaccine within 3 months after receiving study vaccination.
4. After 03 September 2015, any subject who has household contact with infants less than 1 year of age, persons 65 years of age and older, or immunocompromised individuals.

For Phase 1B and Phase 1B Extension:

1. Receipt of seasonal influenza vaccine in the past six months and planned receipt of seasonal influenza vaccine within 3 months after receiving study vaccination.

Specifically Phase 1B Extension:

1. History of medically-attended altered mental status or inner ear (not including hearing loss), labyrinth and cerebellar disorders within 3 months prior to enrollment.
2. Use of concomitant medications that may be nephrotoxic as judged by the investigator.

For Phase 1A, Phase 1B and Phase 1B Extension:

1. Inability to provide informed consent or complete study activities, for example, due to dementia or other impairment.
2. Have an acute illness within 72 hours prior to study vaccination
3. An acute febrile illness within 24 hours prior to vaccination. Vaccination will be deferred until the participant has been afebrile for at least 24 hours.
4. Signs and symptoms of an acute infectious respiratory illness. Vaccination will be deferred until the symptoms resolve.
5. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation.
6. Have immunosuppression as a result of an underlying illness or immunosuppressive treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
7. Have known active neoplastic disease or a history of any hematologic malignancy.
8. Thrombocytopenia or bleeding disorder contraindicating IM vaccination. Receipt of anticoagulants in the three weeks preceding inclusion.
9. Positive screen for HIV, hepatitis B, or hepatitis C infection.
10. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene or squalene-based adjuvants, or other components of the study vaccine.
11. Have a history of severe or life threatening reactions following previous immunization with licensed or unlicensed influenza virus vaccines or a vaccine containing any of the same substances.
12. Have a history of Guillain-Barré Syndrome.
13. Have a history of neuralgia, paresthesia, neuritis, convulsions, or encephalomyelitis within 90 days prior to study vaccination.
14. Have a history of autoimmune disease, including, but not limited to, neuroinflammatory diseases, vasculitis, clotting disorders, dermatitis, arthritis, thyroiditis, or muscle or liver disease.
15. Have a history of kidney disease or use of concomitant nephrotoxic medications.
16. Have a history of alcohol or drug abuse within 5 years prior to study vaccination or drug addiction that may interfere with trial procedures.
17. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
18. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
19. Have taken oral or parenteral corticosteroids of any dose within 30 days prior to study vaccination.
20. Continuous or sporadic use of oral prednisone in the 90 days preceding vaccination.
21. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as >800mcg/day of beclomethasone dipropionate CFC or equivalent.
22. Planned receipt of another vaccine in the four weeks following the trial vaccination.
23. Received any licensed live vaccine within 30 days prior to the study vaccination or planned receipt from the study vaccination through 28 days after the study vaccination.
24. Received any licensed inactivated vaccine within 14 days prior to the study vaccination or planned receipt from the day of study vaccination through 28 days after the study vaccination.
25. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
26. Received an experimental agent within 30 days prior to the study vaccination, or expects to receive an experimental agent, other than from participation in this study, during the study period.
27. Are participating or plan to participate in another clinical trial with an interventional agent during the study period.
28. Plan to travel outside the U.S. (continental U.S., Hawaii and Alaska) within the 28 days following study vaccination.
29. Blood donation within 30 days prior to enrollment and within 30 days after the last blood draw.
30. Personal or family history of narcolepsy with or without cataplexy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with solicited local and systemic AEs | 14 Days after Vaccination
Number of Participants with Late-Onset Local and Systemic AEs | 16 days after Vaccination for the remaining duration of the study
Number of Participants with laboratory abnormalities | 7, 14 and 28 Days after Vaccination
Occurrence of vaccine-related SAEs | Duration of Study
Geometric mean titer (GMT) of hemagglutination inhibition assay (HAI) antibodies | 28 days after Vaccination
Seroconversion rate of HAI antibody titer | 28 days after Vaccination
Geometric mean fold increase (GMFI) of HAI antibodies (post-vaccination titer relative to pre-vaccination titer) | 28, 84, and 168 days after Vaccination

SECONDARY OUTCOMES:
Occurrence of unsolicited AEs related to vaccine | 1 to 14, 15 to 29, and 30 to 85 Days after Vaccination
Occurrence of adverse events of special interest (AESI) | Up to 12 months after Vaccination
Comparison of rates of unsolicited AEs related to vaccine at intervals following vaccination | 1 to 14 days, 15 to 29 days, and 30 to 85 days after Vaccination
Seroprotection rate of HAI antibody titers (proportion of participants with ≥40 reciprocal antibody titer) | 7, 14, 28, 84, and 168 days after Vaccination

OTHER OUTCOMES:
Seroprotection rate of HAI antibody titers (proportion of participants with ≥1:80, 1:160, and 1:320 HAI antibody titer for each of the strains) | 7, 14, 28, 84, and 168 days after Vaccination
GMFI of HAI antibodies | 7 and 14 days after Vaccination
GMT of HAI antibodies to non-vaccine strains of influenza A and B | 28 and 84 days after Vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey J Gorse, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Gorse GJ, Grimes S, Buck H, Mulla H, White P, Hill H, May J, Frey SE, Blackburn P. MAS-1, a novel water-in-oil adjuvant/delivery system, with reduced seasonal influenza vaccine hemagglutinin dose may enhance potency, durability and cross-reactivity of antibody responses in the elderly. Vaccine. 2022 Mar 1;40(10):1472-1482. doi: 10.1016/j.vaccine.2022.01.035. Epub 2022 Feb 4. PMID 35125224
- [Derived] Gorse GJ, Grimes S, Buck H, Mulla H, White P, Hill H, May J, Frey SE, Blackburn P. A phase 1 dose-sparing, randomized clinical trial of seasonal trivalent inactivated influenza vaccine combined with MAS-1, a novel water-in-oil adjuvant/delivery system. Vaccine. 2022 Feb 23;40(9):1271-1281. doi: 10.1016/j.vaccine.2022.01.034. Epub 2022 Feb 4. PMID 35125219